CLINICAL TRIAL: NCT04001218
Title: Neck Pain - Motor and Sensory Aspects
Brief Title: Head Repositioning Accuracy During Experimental Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Associate professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N20120018_Subproject 1d
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Healthy; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the painful condition or the control condition first before crossing over to opposite condition.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painful condition (Experimental): Participants will be injected with 0.5ml hypertonic saline (5.8%) into a neck muscle
  Interventions: Drug: Injection of hypertonic saline
- Control condition (Experimental): Participants will be injected with 0.5ml Isotonic saline (0.9%) into a neck muscle
  Interventions: Drug: Injection of Isotonic saline

INTERVENTIONS:
Drug: Injection of hypertonic saline — Painful condition: Participants will be injected in a neck muscle with 0.5ml of hypertonic saline (5.8%)
  Other Names: Hypertonic saline (5.8%)
  Arms: Painful condition
Drug: Injection of Isotonic saline — Control condition: Participants will be injected in a neck muscle with 0.5ml isotonic saline (0.9%)
  Other Names: Isotonic saline (0.9%)
  Arms: Control condition

SUMMARY:
This study investigates if/how an experimentally applied neck muscle pain influences head repositioning error in healthy participants.

DETAILED DESCRIPTION:
Healthy volunteers will participate in a single session study with a crossover design.

During the study healthy participants will be randomized to either receive a injection of hypertonic saline (painful injection) or isotonic saline (control injection) in a neck muscle.

Head repositioning accuracy will be assessed with and without performing a cognitive task.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-50 years
* Right handed
* Able to speak, read and understand Danish or English
* Normal pain free neck and shoulder range of motion

Exclusion Criteria:

* Pain from the neck or shoulder area
* Prior surgery in neck or shoulder
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Self reported neurologic, musculoskeletal or mental illnesses

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Change in head repositioning accuracy | Within session (session lasts approximately 2 hours)
  Participants will be blindfolded and asked asked to, from a neutral position, to move the head into full range of motion before returning to to a neutral position again. The difference between the start and end position will be used as an estimate of head repositioning error.

SECONDARY OUTCOMES:
Change in perceived pain | Within session (session lasts approximately 2 hours)
  Pain will be scored using a scale from 0-10 with 0 being no pain and 10 being worst imaginable pain, by drawing on body charts and choosing words from the McGill Pain Questionnaire.
Change in perceived performance of head repositioning accuracy test | Within session (session lasts approximately 2 hours)
  Likert scores of the perceived difficultness (0=no problems, 1=minimally difficult, 2=somewhat difficult, 3=fairly difficult, 4= very difficult, 5=unable to perform)

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Dept. Of Health Science and Technology, SMI, Aalborg University, Aalborg, Denmark